CLINICAL TRIAL: NCT06849063
Title: 3D-MRE-Based Evaluation of Biomechanical Heterogeneity in Pancreatic Cancer and Its Clinical Prognosis
Brief Title: Assessment of the Prognosis of Pancreatic Cancer Patients Using 3D MRE
Status: Recruiting | Type: Observational
Sponsor: Yu Shi (Other)
Responsible Party: Sponsor-Investigator, Yu Shi, Associate professor, Shengjing Hospital
Organization: Shengjing Hospital (Other)
Other Study IDs: ShengjingH-chem-PDAC
Record Dates: First submitted 2025-02-23; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer,; Magnetic Resonance Elastography; Prognosis; Biomechanics
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with resectable pancreatic cancer: Investigators anticipate that 150 resectable pancreatic cancer participants are enrolled in this group and all participants undego magnetic resonance imaging
  Interventions: Diagnostic Test: magnetic resonance imaging
- patients with unresectable pancreatic cancer: Investigators anticipate that 50 unresectable pancreatic cancer participants are enrolled in this group and all participants undego magnetic resonance imagin.
  Interventions: Diagnostic Test: magnetic resonance imaging

INTERVENTIONS:
Diagnostic Test: magnetic resonance imaging — all participants undergo novel MR sequences, including 3D MRE#DCE-MRI#IVIM-DWI#T1/T2 mapping.
  Other Names: MR elastrogaphy

SUMMARY:
Pancreatic ductal adenocarcinoma (PDAC), representing 85-95% of pancreatic cancers, is a highly lethal malignancy with a dismal 5-year survival rate below 8%. Emerging evidence highlights the critical need for non-invasive imaging biomarkers to stratify prognosis and guide therapeutic strategies. Notably, the biomechanical properties of PDAC-associated extracellular matrix (ECM), characterized by extensive interstitial fibrosis, are intrinsically linked to tumorigenesis, progression, and metastatic dissemination. Three-dimensional magnetic resonance elastography (3D-MRE), as an advanced imaging modality, enables precise quantification of tissue shear stiffness in both normal pancreatic parenchyma and neoplastic lesions. Significantly, the biomechanical heterogeneity captured by MRE holds untapped potential to serve as a prognostic biomarker for PDAC. Despite its technical merits, no studies to date have systematically explored MRE-derived imaging signatures in predicting PDAC survival outcomes or therapeutic responses, underscoring a pivotal gap in translational oncology research.

DETAILED DESCRIPTION:
Pancreatic ductal adenocarcinoma (PDAC), constituting 85-95% of pancreatic cancers, ranks among the most lethal malignancies globally, with a dismal 5-year survival rate below 8%. Identifying robust prognostic or predictive biomarkers is critical for risk stratification and prospective therapeutic evaluation in clinical trials. The extracellular matrix (ECM) surrounding PDAC is characterized by extensive interstitial fibrosis, a pathological hallmark intrinsically linked to tumor initiation, progression, and metastatic dissemination. While the ECM exerts dual roles in modulating cancer biology through multifaceted mechanisms, compelling experimental evidence confirms that ECM stiffening in PDAC accelerates tumor aggressiveness and correlates significantly with reduced patient survival. Noninvasive quantification of tumor mechanical properties (e.g., stiffness) prior to treatment could provide critical insights into tumor biology, prognostic stratification, and personalized therapeutic decision-making.

Advanced three-dimensional magnetic resonance elastography (3D-MRE) enables precise, noninvasive mapping of shear stiffness across both healthy pancreatic tissue and neoplastic lesions. Despite its technical promise, the translational potential of MRE-derived imaging biomarkers for predicting PDAC prognosis remains unexplored, with no systematic studies reported domestically or internationally to date.

ELIGIBILITY:
Inclusion Criteria:

1. granting of written informed consent
2. age ≥18 years
3. no history of extrapancreatic malignancy
4. no preoperative biliary drainage
5. definitive histologic evidence of PDAC in excisional biopsy
6. with no less than three months of postoperative mortality or six months of follow- up

Exclusion Criteria:

1. inability to re-review of tissue specimens
2. unacceptable estimates of MRE parameters, specifically invalid wave data during postprocessing, inconsistent breath-holdings, intolerable pain, and MRE hardware disconnection
3. tumor diameters <1.0 cm
4. withdrawal/dropout during follow-up

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: participants aged 18-80 years
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Analyzing the measurement accuracy of MRE. | 9 months
  The hardness was measured by a hardness tester during the operation, and the mechanical parameters were measured by atomic force microscopy of the in vitro specimen. The measurement accuracy of MRE was analyzed by comparing the hardness tester and atomic force microscope results.
Radiological assessment of tumor stiffness | 9 months
  A self-written script program in MATLAB is used to read and analyze mechanical group diagrams and waveform diagrams in three directions of x, y, and z, and a region of interest (ROI) delineation function is embedded. After drawing the ROI, an Excel file containing the corresponding values is automatically generated, and the average values of various mechanical parameters are calculated, including shear modulus (|G*|, SS), storage modulus (G', SM), loss modulus (G'', LM) and damping ratio (#, DR).
Evaluation of tumor response to chemotherapy. | 12 months
  RECIST criteria (version 1.1) were used to objectively evaluate the response to chemotherapy.
Investigating the correlation between magnetic resonance elastography (MRE) shear stiffness and clinical outcomes in pancreatic cancer patients. | 9 months
  Optimize longitudinal follow-up for pancreatic cancer patient subgroups. Utilizing shear stiffness measurements from magnetic resonance elastography (MRE) and clinical outcomes among distinct patient groups, generate Kaplan-Meier survival curves to determine the clinical utility of biomechanical characterization in prognosticating pancreatic cancer. Statistical analyses were conducted with R and GraphPad Prism.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Shi, MD.PhD., Principal Investigator — Study Principal Investigator
Locations (1):
- Shengjing hospital of China medical university, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No